CLINICAL TRIAL: NCT04742634
Title: A Phase I/II Trial of Pre-emptive Therapy With DEC-C to Improve Outcomes in MDS Patients With Measurable Residual Disease Post Allogeneic Hematopoietic Cell Transplant
Brief Title: Pre-emptive Therapy With DEC-C to Improve Outcomes in MDS Patients With Measurable Residual Disease Post Allogeneic Hematopoietic Cell Transplant
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202103255
Record Dates: First submitted 2021-01-28; First posted 2021-02-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Phase I Dose Level 1: DEC-C (Experimental): * Bone marrow biopsy & MyeloSeq-HD will be obtained on Day 30 post-transplant. MRD positivity is defined as the presence of at least one somatically acquired mutation detected prior to transplant that persists at Day 30 post-transplant with a variant allele frequency of ≥ 0.2%. MRD-positive patients will receive up to 5 cycles of DEC-C prior to the Day 180 bone marrow evaluation. If the Day 180 MyeloSeq-HD shows that MRD is still detectable in the opinion of the MGI board-certified molecular pathologist but below 0.5% and patient has tolerated initial treatment without toxicity, the patient may continue treatment. If it shows a lack of MRD, the patient will be moved to the post-treatment surveillance arm. If it shows any mutation detection prior to transplant that persists with a variant allele frequency of ≥ 0.2%VAF, the patient will receive up to an additional 6 cycles of DEC-C.
  * 35 mg decitabine/100 mg cedazuridine taken by mouth once daily on Days 1, 2, 3 of a 28 day cycle.
  Interventions: Drug: DEC-C; Device: MyeloSeq-HD
- Phase I Dose Level 2: DEC-C (Experimental): * Bone marrow biopsy & MyeloSeq-HD will be obtained on Day 30 post-transplant. MRD positivity is defined as the presence of at least one somatically acquired mutation detected prior to transplant that persists at Day 30 post-transplant with a variant allele frequency of ≥ 0.2%. MRD-positive patients will receive up to 5 cycles of DEC-C prior to the Day 180 bone marrow evaluation. If the Day 180 MyeloSeq-HD shows that MRD is still detectable in the opinion of the MGI board-certified molecular pathologist but below 0.5% and patient has tolerated initial treatment without toxicity, the patient may continue treatment. If it shows a lack of MRD, the patient will be moved to the post-treatment surveillance arm. If it shows any mutation detection prior to transplant that persists with a variant allele frequency of ≥ 0.2%VAF, the patient will receive up to an additional 6 cycles of DEC-C.
  * 35 mg decitabine/100 mg cedazuridine taken by mouth once daily on Days 1-4 of a 28 day cycle.
  Interventions: Drug: DEC-C; Device: MyeloSeq-HD
- Phase II MRD Positive: DEC-C (Experimental): * 35 mg decitabine/100 mg cedazuridine taken by mouth once daily per the schedule determined in the Phase I portion of the study. Cycle 1 Day 1 may take place between Day 42 and Day 100 post-transplant. MRD-positive patients will receive up to 5 cycles of DEC-C prior to the Day 180 bone marrow evaluation.
  * Bone marrow biopsy with MyeloSeq-HD will be obtained on Day 180 post-transplant. If the Day 180 MyeloSeq-HD shows that MRD is still detectable in the opinion of the MGI board-certified molecular pathologist but below 0.5% and patient has tolerated initial treatment without toxicity, the patient may continue treatment. If it shows a lack of MRD, the patient will be moved to the post-treatment surveillance arm. If it shows any mutation detection prior to transplant that persists with a variant allele frequency of ≥ 0.2%VAF, the patient will receive up to an additional 6 cycles of DEC-C.
  Interventions: Drug: DEC-C; Device: MyeloSeq-HD
- Phase II MRD Negative: Observation Arm (Active Comparator): * In phase II, up to 77 patients who do not have MRD positivity on Day 30 post-transplant (i.e., the absence of at least one somatically acquired mutation detected prior to transplant that persists at Day 30 post-transplant with a variant allele frequency of ≥ 0.2%) will be placed on the observation arm and treated with standard of care.
  * Patients on the observation arm will be followed every 3 months for 2 years and every 6 months for 3 years for progression and survival
  Interventions: Device: MyeloSeq-HD

INTERVENTIONS:
Drug: DEC-C — * DEC-C will be provided by Taiho Pharmaceuticals.
  * Cycle 1 Day 1 may take place between Day 42 & Day 100 post-transplant.
  Other Names: decitabine + cedazuridine; ASTX727; INQOVI®
  Arms: Phase I Dose Level 1: DEC-C; Phase I Dose Level 2: DEC-C; Phase II MRD Positive: DEC-C
Device: MyeloSeq-HD — -Laboratory test developed at Washington University School of Medicine

SUMMARY:
The investigators hypothesize that early measurable residual disease (MRD)-guided pre-emptive therapy with decitabine + cedazaridine (DEC-C) will decrease the risk of progression in post-transplant myelodysplastic syndromes (MDS) patients with persistent mutations (molecular MRD). To detect molecular MRD, the investigators will perform ultra-deep, error-corrected panel-based sequencing (MyeloSeq-HD) at Day 30 in post-transplant MDS patients. The investigators will treat patients with detectable molecular MRD with DEC-C to determine if pre-emptive, MRD-guided therapy with DEC-C decreases relapse rates and improves progression-free survival.

ELIGIBILITY:
This study uses a two-stage eligibility process. Step 1 assesses eligibility prior to the MyeloSeq-HD assay being performed, while Step 2 assesses eligibility of MRD-positive patients for the intervention arm and MRD-negative patients for the observation arm. Patients who are MRD-positive who are determined to be ineligible to continue into the intervention arm must satisfy the eligibility criteria for the observation arm in order to be enrolled in that arm.

Eligibility Criteria for MyeloSeq-HD Assay (Step 1)

* Diagnosis of myelodysplastic syndromes (MDS) based on World Health Organization classification (2016 revision) who have received an allogeneic hematopoietic cell transplant. Any stem cell source, conditioning regimen, and immunosuppression regimen as determined by the treating physician, per institutional guidelines, is permitted. Patients may have received any therapy, or no therapy, prior to transplant.
* 18 to 75 years of age.
* Must have undergone gene panel testing prior to the start of transplant conditioning and must have at least one somatically acquired mutation that is interrogated by the MyeloSeq-HD panel. If the patient has a variant that is known to be a germline/inherited myeloid predisposition gene in that patient, this variant cannot and will not be used as evidence of MRD positivity. If the pre-transplant gene panel testing is a next-generation sequencing panel other than the MyeloSeq platform, the outside report will be reviewed by the PI and the molecular pathologists at the McDonnell Genome Institute to ensure eligibility.
* Willing to comply with the treatment assignment:

  * Intent to proceed with DEC-C therapy if one or more variants detected prior to transplant persists at Day 30 post-transplant with a variant allele frequency of ≥ 0.2%.
  * Intent to proceed with standard of care as determined by the treating physician on the observation arm (no DEC-C intervention) if no variants detected prior to transplant persist at Day 30 post-transplant with a variant allele frequency of ≥ 0.2%, or if the other inclusion criteria are not met.
* Not currently receiving any investigational agents.
* Ability to understand and willingness to sign an IRB-approved written informed consent document (or that of legally authorized representative, if applicable).

Eligibility Criteria for Step 2 Step 2A Inclusion Criteria (DEC-C Intervention Arm)

* One or more somatically acquired variants that were present prior to transplant detected by the MyeloSeq-HD panel at Day 30 post-transplant, with a variant allele frequency of ≥ 0.2%
* Within Days 42-100 post-transplant.
* ≤ 5 % bone marrow myeloblasts on the Day 30 post-transplant biopsy.
* Absolute neutrophil count (ANC) ≥ 1.0 X 109/L and platelets ≥ 50 X 109/L.
* Only patients with adequately controlled GVHD ≤ Grade 2 are eligible for the DEC-C intervention arm. Patients with active grade 3 or higher GVHD are ineligible for the DEC-C intervention arm.
* ECOG performance status ≤ 2
* Adequate renal and hepatic function as described below:

  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 IULN
  * Creatinine clearance ≥ 30 mL/min using Cockcroft-Gault Formula below:

CrCl = [(140-age) x body weight in kg]/(serum creatinine in mg/dL x 72) x 0.85 if female

*NOTE: If, in the opinion of the treating physician, bilirubin is elevated secondary to hemolysis or Gilbert's disease, the patient may be eligible after discussion with the Washington University PI

* Decitabine has been shown to be teratogenic in animal studies and use of IV decitabine in the first trimester of pregnancy has been associated with major birth defects. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men and women treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 6 months after completion of the study.

Step 2B Inclusion Criteria (Observation Arm)

* EITHER ≤ 5 % bone marrow myeloblasts on the Day 30 post-transplant biopsy OR enrolled in the study with > 5% bone marrow myeloblasts on the Day 30 post-transplant biopsy but not meeting eligibility criteria for the intervention arm.
* Not receiving any investigational agents.

Step 2A Exclusion Criteria

* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to DEC-C or other agents used in the study.
* Concomitant administration of drugs metabolized by cytidine deaminase
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum/urine pregnancy test no more than 10 days prior of the start of the first cycle of DEC-C.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2033-11-30 (Estimated); Study Completion 2033-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicities (Phase I only) | Completion of cycle 1 (each cycle is 28 days) for all phase I participants (estimated to be 13 months)
  -Dose-limiting toxicities (DLTs) are defined as any of the following adverse events that occur during the DLT observation period (Cycle 1) during the phase I portion of the study, determined to be possibly, probably, or definitely related to the study drug:
  * Grade 4 neutropenia or grade 4 thrombocytopenia in the absence of increased blasts and/or evidence of persistent MDS at the end of Cycle 1.
  * Any grade 3 or higher non-hematologic toxicity except for grade 3 vomiting or diarrhea not requiring tube feeding, total parenteral nutrition, or requiring or prolonging hospitalization, or grade 3 or 4 isolated electrolyte abnormalities that last <72 hours.
  * Any other non-hematologic toxicity that is clinically significant and/or unacceptable that does not respond to supportive care, results in disruption of dosing schedule more than 28 days, or is judged to be a DLT by the Investigator.
  * Confirmed Hy's law cases will be considered a DLT
Maximum tolerated dose (MTD) (Phase I only) | Completion of cycle 1 (each cycle is 28 days) for all phase I participants (estimated to be 13 months)
  -The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which ≥ 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle.
Recommended phase II dose (Phase I only) | Completion of cycle 1 (each cycle is 28 days) for all phase I participants (estimated to be 13 months)
  -The recommended phase II dose will be less than or equal to the maximum tolerated dose
Progression-free survival (PFS) (Phase II recommended dose only) | 1 year post-transplant
  -Progression-free survival: Defined as the interval from the date of transplant to disease progression or death, whichever is first. Patients without documented disease progression or death at the time of analysis will be censored at the date of last adequate tumor assessment.
Rate of relapse (Phase II recommended dose only) | 1 year post-transplant
  -Disease progression/relapse post-transplant is defined as >5% myeloblasts in the bone marrow, evidence of extramedullary disease, reemergence of pre-transplant cytogenetic abnormalities, or intervention by the treating physician (such as withdrawal of immunosuppression) for reemergence of pre-transplantation morphologic abnormalities that are likely relapsed disease in the opinion of the treating physician. Censoring rules for the Relapse endpoint include: Patients who do not relapse will be censored at the date of last disease assessment where no relapse was documented; Patients who die without relapse will be censored at the date of death if no relapse was observed prior to death. Patients who withdraw consent or are lost to follow-up will be censored at the date of last disease assessment showing no evidence of relapse; Patients who start a new anti-cancer therapy before documented relapse will be censored at the date of last disease assessment before the start of the new therapy.

SECONDARY OUTCOMES:
Overall survival (OS) (Phase II recommended dose only) | 1 year post-transplant
  -Overall survival: Defined as the date of transplant to the date of death from any cause. Patients still alive at the time of analysis will be censored at the date they were last known to be alive.
Percentage of patients requiring DEC-C dose adjustment/delay (Phase II recommended dose only) | Through completion of treatment (estimated to be 168 days)
Percentage of cycles given on time/at dose (Phase II recommended dose only) | Through completion of treatment (estimated to be 168 days)
Change in mutational MRD disease burden as measured by variant allele frequency (VAF) (Phase II recommended dose only) | Day 180
  -In patients who have at least 1 cycle of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Meagan Jacoby, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results in the article, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months after publication.
Access Criteria: Anyone who wishes to access the data. Please email principal investigator.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu